CLINICAL TRIAL: NCT03747796
Title: Evaluation of the Impact of Semi-sitting Position Versus Supine Position on Gastric Emptying in Children Using Gastric Ultrasound: a Randomized Controlled Trial
Brief Title: The Impact of Semi-sitting Position Versus Supine Position on Gastric Emptying in Children Using Gastric Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor of anesthesia and critical care, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-92-2018
Record Dates: First submitted 2018-11-17; First posted 2018-11-20 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia; Fasting
MeSH Terms: conditions — Fasting | interventions — Supine Position

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supine position (Active Comparator): The children will be in the supine position after ingestion of a standard volume of clear fluid.
  Interventions: Other: Supine position
- Semi-sitting position (Experimental): The children will be in the semi-sitting position after ingestion of a standard volume of clear fluid.
  Interventions: Other: Semi-sitting position

INTERVENTIONS:
Other: Supine position — The children will be placed in the supine position after ingestion of a standard volume of clear fluid
  Arms: supine position
Other: Semi-sitting position — The children will be placed in the semi-sitting position after ingestion of a standard volume of clear fluid
  Arms: Semi-sitting position

SUMMARY:
The aim of this work is to evaluate the effect of semi sitting versus supine positions on gastric emptying of fluids in children using gastric ultrasound.

The investigators hypothesize that gastric emptying in children might be faster if the patient is in semi-sitting position. This hypothesis could impact the current guidelines for peri-operative fasting. Moreover, if this proved effective, could be used for enhancement of gastric emptying before emergency operations in non-fasting patient.

DETAILED DESCRIPTION:
Dealing with preoperative fasting requires a meticulous balance ensuring patient safety and lessening patient's discomfort. Although fasting is a basic requirement for avoiding pulmonary aspiration, it is sometimes associated with patient discomfort and hypoglycemia. According to the current guidelines for preoperative fasting of children, fasting is required for 2-hours, 4-hours, and 6-hours period after ingestion of water, breast milk, and infant formula respectively. Limited data is available for the effect of patient positioning on gastric emptying. A previous study had reported that gastric emptying of non-nutrient liquids was faster in the sitting position compared with the left lateral position . Another study showed similar findings after nutritive liquid and solid meals; whilst, a third study had reported that gravity has a little effect on gastric emptying.

In pediatric population the effect of posture on the duration of gastric emptying is not well investigated.

Gastric ultrasound is a valid, accurate, reproducible, non-invasive, bedside test for evaluation of the gastric volume. gastric ultrasound has been validated in adults as well as children for estimating the volume of gastric contents and evaluating gastric emptying.

The aim of this work is to evaluate the effect of semi sitting versus supine positions on gastric emptying of fluids in children using gastric ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Children 4 to 16 years of age.
* Fasting for elective surgery.

Exclusion Criteria:

* Gastrointestinal problems that may delay gastric emptying.
* Recent abdominal operations.
* Major systemic diseases which could impact gastric emptying.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-13 (Actual)

PRIMARY OUTCOMES:
Number of children who have complete gastric emptying | 30 minutes after ingestion of clear fluid
  Number of children who have complete gastric emptying defined as return of the antral cross-sectional area to the baseline reading

SECONDARY OUTCOMES:
Antral cross-sectional area corrected to the body weight | 3 hours after ingestion of clear fluid
  Antral cross-sectional area divided by the body weight
Hunger satiety score | 3 hours after ingestion of clear fluid
  A score which measures the degree of patient satiety. The score ranges from zero which is the worst value, to five which is the best value.
Number of children who have complete gastric emptying | 60 minutes after ingestion of clear fluid
  Number of children who have complete gastric emptying after 60 minutes, defined as return of the antral cross-sectional area to the baseline reading
Number of children who have complete gastric emptying | 120 minutes after ingestion of clear fluid
  Number of children who have complete gastric emptying after 120 minutes, defined as return of the antral cross-sectional area to the baseline reading

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Rady, Professor, Study Director — Cairo University
Locations (1):
- Ahmed Mohamed Hasanin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No